CLINICAL TRIAL: NCT00072592
Title: An Open Label Pilot Study Examining the Use of Rituximab in Patients With Wegener's Granulomatosis Who Have Experienced Disease Relapse on Standard Therapies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040022; 04-I-0022
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Wegener's Granulomatosis
Keywords: ANCA; B Lymphocyte; Vasculitis; Treatment; Remission; Wegener Granulomatosis; WG
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Vasculitis | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This study will examine the use of rituximab in patients with Wegener's granulomatosis (WG) who have experienced a relapse of the disease through standard therapies. Rituximab is an antibody directed against the human protein called CD20, found on the surface of normal and abnormal B lymphocytes. Rituximab decreases the number of B lymphocytes. This study will examine the safety of rituximab in WG and rituximab's ability to reduce the level of circulating antineutrophil cytoplasmic antibodies (ANCA), which are antibodies that react to substances found in white blood cells. ANCA have been found to be strongly associated with WG. The study will also explore whether rituximab can reduce the occurrence of disease relapse. WG is a disease marked by inflammation of blood vessels. It can involve many different parts of the body, including the sinuses, lungs, kidneys, brain, nerves, eyes, intestinal tract, skin, joint, heart, and others. Before the use of cytotoxic drug therapy, WG was almost always fatal if untreated, with a mortality rate of 93% within 2 years.

Patients 18 to 75 years of age who have a history of at least one relapse of the disease despite standard treatments, who have had active WG within the previous 12 months and are in remission, who are receiving either methotrexate or azathioprine for remission maintenance, and who have circulating ANCA, may be eligible for this study.

A minimum of 22 visits to the clinic will be required to complete the entire study. Patients will undergo a comprehensive medical evaluation, with laboratory studies and x-rays. There may also be consultations and possible biopsies of affected organs only if medically indicated for diagnosis and treatment of the disease. In the 4-week period that patients will receive rituximab infusions, the methotrexate or azathioprine will be continued at the same dosage unless there are side effects that requite the medication to be temporarily stopped or the dosage reduced. Patients will receive four doses of rituximab, at 375 mg per meter squared of body surface area, once a week. It will be infused into a vein, through an intravenous catheter. For the first dose, patients will be admitted as inpatients for at least 24 hours, for monitoring during the infusion and for any reactions associated with it. The second, third, and fourth rituximab infusions may be given either on an inpatient or outpatient basis to be decided on how the patient tolerates the first infusion.

Following the four infusions, there will be blood tests to monitor the safety of the medication and the status of the disease, to be done at home every week for 4 weeks. Results will be sent to the researchers by fax. Patients will be asked to return to the clinic 1 month after the fourth infusion and every 1 to 3 months afterward. If there are no side effects or a relapse of the disease, the methotrexate or azathioprine will be continued for 2 years past remission. If by then the disease then remains in remission, the dose of either medication will be gradually decreased and eventually stopped. The usual schedule is to reduce methotrexate by 2.5 mg per month and to reduce azathioprine by 25 mg per month. If at that point there are no signs of active disease, the patients' illness will be considered to be in continued remission and no further treatment will be necessary. If relapse does occur, treatment would be different than previously. In most cases, treatment would involve prednisone and cyclophosphamide or methotrexate If the ANCA finding is negative after rituximab treatment and again becomes positive, and there is evidence of a return of B lymphocytes, patients may receive a second course of four rituximab infusions.

DETAILED DESCRIPTION:
This pilot study will seek to investigate the use of rituximab in patients with Wegener's granulomatosis who have experienced disease relapse through standard therapies. Rituximab is a chimeric monoclonal antibody directed against CD20, which induces B cell death and results in rapid and sustained depletion of circulating and tissue-based B cells. The objectives of this protocol will be to establish the safety of rituximab in Wegener's granulomatosis, to examine the ability of rituximab to reduce the level of circulating antineutrophil cytoplasmic antibodies (ANCA), and to preliminarily explore whether rituximab is able to prevent disease relapse. This prospective standardized open label trial will enroll 10 patients who have a well-documented history of disease relapse while receiving immunosuppressive therapy given according to published regimens and who are ANCA positive after remission induction. Patients will be enrolled once they have achieved remission from a recent relapse and are receiving either methotrexate or azathioprine for remission maintenance. All patients will receive rituximab 375 mg/M(2) once a week for 4 weeks. During and following the rituximab treatment period, patients will remain on their remission maintenance agent of methotrexate or azathioprine. Patients who are enrolled while on prednisone will continue to taper the dosage to discontinuation as medically permitted. Following the 4 weekly infusions of rituximab, patients will be followed prospectively for evidence of effective B cell depletion, features of drug toxicity, level of circulating ANCA, and clinical disease status. Patients whose ANCA levels become undetectable following the infusion of rituximab may be retreated with a second 4 week course of rituximab should their ANCA titer become positive (greater than or equal to 1:40) and there has been a return of B cells in the peripheral blood. Methotrexate or azathioprine will be continued for two years past remission, after which time, this will be tapered and discontinued. Patients will continue to be monitored for two years off all immunosuppressive therapy or if a disease relapse should occur, for a minimum of 12 months after the last rituximab infusion.

ELIGIBILITY:
INCLUSION CRITERIA:

Documentation of WG based on clinical characteristics and histopathologic and/or angiographic evidence of vasculitis. In the absence of histopathologic and/or angiographic evidence of vasculitis, patients who meet one of the following criteria and in whom infectious and autoimmune diseases that may mimic WG have been excluded will also be eligible:

A positive assay for anti-PR-3 or anti-MPO autoantibodies (ANCA) and the presence of glomerulonephritis defined by red blood cell casts and proteinuria or renal biopsy showing necrotizing glomerulonephritis in the absence of immune deposits.

A positive assay for anti-PR-3 or anti-MPO autoantibodies and at least 2 of the following: the presence of granulomatous inflammation on biopsy; abnormal chest radiograph (defined as the presence of nodules, fixed infiltrates, or cavities); nasal/oral inflammation on clinical examination.

Age 18-75 years.

Previous history of greater than or equal to 1 disease relapse as defined in Appendix I in patients fitting one of the below categories:

Disease relapse occurred while receiving MTX or AZA for remission maintenance following remission induction with daily CYC according to standard regimens on which there has been published data

Disease relapse occurred while on MTX following MTX induction according to the standard regimen on which there has been published data (98) in a patient who is unable to receive or is intolerant to daily CYC.

Active WG within the past 12 months for which the patient received induction therapy with glucocorticoids combined with daily CYC or MTX according to standard regimens

Evidence of current disease remission as defined in Appendix I and is currently receiving remission maintenance therapy consisting of MTX or AZA according to standard regimens. Patients may concurrently be receiving prednisone that is being tapered. Patients who completed their prednisone taper and are no longer receiving systemic glucocorticoids will be eligible if they are within 6 months of the time of prednisone discontinuation.

Circulating ANCA as defined by the presence of antibodies detectable by indirect immunofluorescence performed by the NIH Clinical Immunology laboratory at a titer of greater than or equal to 1:40 on two determinations done at least 4 weeks apart. Patients who are historically ANCA positive and become ANCA negative during remission induction will be eligible if they again become positive to a level of greater than or equal to 1:40 on two determinations done at least 4 weeks apart at a prednisone dose of less than or equal to 50mg QOD or within 6 months following the discontinuation of prednisone.

Willingness to travel to the NIH

Willingness of both women and men to use an effective means of birth control while receiving treatment through this study. Effective contraception methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap or sponge, or hormonal contraception.

EXCLUSION CRITERIA:

Evidence of active infection, which, in the judgment of the investigator, is of greater danger to the patient than the underlying vasculitis.

Patients who are pregnant or who are nursing infants will not be eligible. Women of childbearing potential must have a negative pregnancy test within one week prior to study entry.

Serological evidence of infection with human immunodeficiency virus (HIV), hepatitis C, or a positive hepatitis B surface antigen. A serological determination will be performed within two weeks of beginning study participation.

Inability to comply with study guidelines.

Hemocytopenia: platelet count greater than 80,000/mm(3), absolute neutrophil count less than 1500/mm(3), hematocrit less than 20% (in the absence of gastrointestinal bleeding or hemolytic anemia).

Known allergy to murine proteins

Use of illegal drugs or alcohol abuse (alcohol use that would prevent a patient from fulfilling the study requirements or that would increase the risk of study procedures.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2003-10; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hoffman GS, Kerr GS, Leavitt RY, Hallahan CW, Lebovics RS, Travis WD, Rottem M, Fauci AS. Wegener granulomatosis: an analysis of 158 patients. Ann Intern Med. 1992 Mar 15;116(6):488-98. doi: 10.7326/0003-4819-116-6-488. PMID 1739240
- [Background] Reinhold-Keller E, Beuge N, Latza U, de Groot K, Rudert H, Nolle B, Heller M, Gross WL. An interdisciplinary approach to the care of patients with Wegener's granulomatosis: long-term outcome in 155 patients. Arthritis Rheum. 2000 May;43(5):1021-32. doi: 10.1002/1529-0131(200005)43:53.0.CO;2-J. PMID 10817555
- [Background] Talar-Williams C, Hijazi YM, Walther MM, Linehan WM, Hallahan CW, Lubensky I, Kerr GS, Hoffman GS, Fauci AS, Sneller MC. Cyclophosphamide-induced cystitis and bladder cancer in patients with Wegener granulomatosis. Ann Intern Med. 1996 Mar 1;124(5):477-84. doi: 10.7326/0003-4819-124-5-199603010-00003. PMID 8602705